CLINICAL TRIAL: NCT01906801
Title: Clinical Efficacy of Glucosamine Plus Diacerein Versus Mono-therapy of Glucosamine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Jatupon Kongtharvonskul, Section for Clinical Epidemiology and Biostatistics, Faculty of Medicine Ramathibodi Hospital, Bangkok, Thailand, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04-56-25
Record Dates: First submitted 2013-07-20; First posted 2013-07-24 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Osteoarthritis; Glucosamine; Diacerein
Keywords: Osteoarthritis; Glucosamine sulfate; Diacerein; Randomized controlled trial
MeSH Terms: conditions — Osteoarthritis | interventions — Glucosamine; diacerein

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glucosamine sulfate & Diacerein (Experimental): Glucosamine sulfate (sachet) 1500 mg and Diacerein 50 mg tablet by mouth once daily for 24 weeks
  Interventions: Drug: Glucosamine sulfate; Drug: Diacerein
- Glucosamine sulfate & Placebo (Active Comparator): Glucosamine sulfate 1500 mg and Placebo (for Diacerein) 50 mg by mouth once daily for 24 weeks
  Interventions: Drug: Glucosamine sulfate; Drug: Placebo (for Diacerein)

INTERVENTIONS:
Drug: Glucosamine sulfate
  Other Names: Viatril-S
Drug: Diacerein
  Other Names: Artrodar
  Arms: Glucosamine sulfate & Diacerein
Drug: Placebo (for Diacerein) — Sugar pill manufactured to mimic Diacerein 50 mg tablet
  Arms: Glucosamine sulfate & Placebo

SUMMARY:
The purpose of this study is to compare pain scores, WOMAC total and subscores, actual and change of joint space width and the rate of gastrointestinal side effects at 4, 8, 12, and 24 weeks between dual-therapy of diacerein and glucosamine versus a mono-therapy of glucosamine in OA patients

ELIGIBILITY:
Adult patients age 50 years or older who have been diagnosed as primary or secondary osteoarthritis of the knee base on clinical criteria of American College of Rheumatology

Inclusion Criteria:

* Clinical diagnosis of primary osteoarthritis
* Mild deformity Clinical (having no varus or valgus deformity, no crepitus) ? Physical examination grade 0 assessed by stress test Radiographic assessment (Kellgrane-lawrance type II-III), a minimum baseline medial tibiofemoral JSW of _2 mm.
* Willing to participate and provide written informed consent

Exclusion Criteria:

* Non-secondary osteoarthritis Rheumatoid arthritis, inflammatory arthritis (e.g. SLE, Gout), post traumatic osteoarthritis, those who received intra-articular treatment of the signal joint with any product (corticosteroids in the previous 2 months, or glycosaminoglycans/hyaluronic acid in the previous 6 months) or had undergone joint lavage andarthroscopic procedures in the previous 6 months.
* No contraindication of using diacerein and glucosamine
* Non-current or ex-users of oral SYSADOA (e.g., glucosamine sulphate, chondroitin sulphate, diacerein, piascledine), anti-depressants, tranquillisers, antacids or antibiotics known hypersensitivity to diacerein, to similar compounds, to the excipients or to paracetamol

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2013-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
pain visual analog scores | 24 weeks

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis (WOMAC) scores | 24 weeks
actual and change of joint space width | 24 weeks
Rate of gastrointestinal side effects | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patarawan Woratanarat, MD, Ph.D, Study Director — Department of Orthopaedics, Faculty of Medicine Ramathibodi Hospital, Bangkok, Mahidol University, Thailand.; Ammarin Thakkinstian, Ph.D, Study Chair — Section for Clinical Epidemiology and Biostatistics, Faculty of Medicine Ramathibodi Hospital, Bangkok, Thailand
Locations (1):
- Department of Orthopaedics, Faculty of Medicine Ramathibodi Hospital, Bangkok, Mahidol University, Bangkok, Thailand

REFERENCES:
- [Derived] Kongtharvonskul J, Woratanarat P, McEvoy M, Attia J, Wongsak S, Kawinwonggowit V, Thakkinstian A. Efficacy of glucosamine plus diacerein versus monotherapy of glucosamine: a double-blind, parallel randomized clinical trial. Arthritis Res Ther. 2016 Oct 12;18(1):233. doi: 10.1186/s13075-016-1124-9. PMID 27729073